CLINICAL TRIAL: NCT00772070
Title: Antibody Responses to a Reduced Dose of Menomune® in Children Who Previously Received an Experimental Tetravalent (A, C, Y, and W-135) Meningococcal Diphtheria Toxoid Conjugate Vaccine, TetraMenD
Brief Title: Study of Reduced Dose of Menomune® in Children Who Previously Received Meningococcal Diphtheria Toxoid Conjugate Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MTA17
Record Dates: First submitted 2008-10-13; First posted 2008-10-15 (Estimated); Results first posted 2009-05-14 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-01

CONDITIONS: Meningitis; Meningococcemia; Neisseria Meningitidis
Keywords: Menactra®; Menomune®; Meningitis; Meningococcemia; Neisseria meningitidis
MeSH Terms: conditions — Meningitis; Meningococcal Infections | interventions — Meningococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Previously received TetraMenD (Experimental): Participants previously received one dose of a Meningococcal vaccine, TetraMenD in Study 603-02.
  Interventions: Biological: A/C/Y/W-135, Meningococcal Polysaccharide Vaccine (Menomune®)
- Meningococcal vaccine-naїve (Experimental): Participants have never received a Meningococcal vaccine in the past.
  Interventions: Biological: A/C/Y/W-135, Meningococcal Polysaccharide Vaccine (Menomune®)

INTERVENTIONS:
Biological: A/C/Y/W-135, Meningococcal Polysaccharide Vaccine (Menomune®) — 0.05 mL, Subcutaneous
  Other Names: Menomune®
  Arms: Previously received TetraMenD
Biological: A/C/Y/W-135, Meningococcal Polysaccharide Vaccine (Menomune®) — 0.05 mL, Subcutaneous
  Other Names: Menomune®
  Arms: Meningococcal vaccine-naїve

SUMMARY:
This study was designed to simulate meningococcal challenge by vaccination with a fractional combined dose of unconjugated meningococcal polysaccharides A, C, Y, and W-135, Menomune® in children who were vaccinated with one dose of TetraMenD at least 18 months earlier.

Primary Objective:

To evaluate and compare the antibody responses to a reduced dose of Menomune® in participants who had previously received a tetravalent meningococcal diphtheria toxoid conjugate vaccine to those responses in participants who received the same reduced dose of Menomune® but had not previously received any meningococcal vaccine.

DETAILED DESCRIPTION:
This was a two stage, controlled, open-label trial. Stage I of the trial simulated meningococcal challenge Stage II of the trial evaluated the meningococcal vaccine naïve participants from Stage I, who had also received a reduced dose of Menomune® vaccine in Stage I and were administered a full dose of Menactra® vaccine 6 months later.

ELIGIBILITY:
Inclusion Criteria :

* Stage I
* Participant is healthy, as determined by medical history and physical examination.
* Participant is at least 3 years of age but not yet 6 years of age at the enrolment.
* For the TetraMenD group: received one dose of TetraMenD as a participant in trial 603-02 no less than 18 months prior to enrolment
* For the Control group: no previous history of any meningococcal vaccination
* Parent/Guardian has signed Institutional Review Board- (IRB-) approved informed consent form.
* Stage II
* Participant is healthy, as determined by medical history and physical examination.
* Participant is at least 3 years of age but not yet 6 years of age at the time of enrollment in Stage 1.
* Enrolled in the Control group only and received one dose of the reduced dose Menomune at Stage 1.
* Parent/Guardian has signed Institutional Review Board- (IRB-) approved informed consent form.

Exclusion Criteria :

* Serious chronic disease (i.e., cardiac, renal, neurologic, metabolic, rheumatologic, psychiatric etc.)
* Known or suspected impairment of immunologic function
* Acute medical illness with or without fever within the last 72 hours or an axillary temperature (≥ 99.5ºF [≥ 37.5ºC]) at the time of inclusion
* For Stage I, history of documented invasive meningococcal disease or previous meningococcal vaccination with exception of those participants recruited from Trial 603-02.
* For Stage II, history of documented invasive meningococcal disease or participant did not receive Reduced-dose Menomune® six months prior.
* Administration of immune globulin, other blood products within the last three months, injected or oral corticosteroids or other immunomodulatory therapy within six weeks of the study vaccine. Individuals on a tapering dose schedule of oral steroids lasting < 7 days may be included in the trial as long as they have not received more than one course within the last two weeks prior to enrollment.
* Antibiotic therapy within the 72 hours prior to vaccination or antibiotic therapy within the 72 hours prior to having any blood sample drawn
* Received any vaccine in the 28-day period prior to study vaccination, or scheduled to receive any vaccination during the 28-day period after study vaccination in Stage 1 of the trial.
* Suspected or known hypersensitivity to any of the vaccine components
* Unavailable for the entire study period or unable to attend the scheduled visits or to comply with the study procedures
* Enrolled in another clinical trial
* Any condition, which, in the opinion of the investigator, would pose a health risk to the participant or interfere with the evaluation of the vaccine.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 173 (Actual)
Dates: Start 2003-03; Primary Completion 2003-08 (Actual); Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (8):
- United States (8):
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Woburn, Massachusetts
  - Bridgeton, Missouri
  - Rochester, New York
  - Pittsburgh, Pennsylvania
  - Sellersville, Pennsylvania
  - Norfolk, Virginia

REFERENCES:
- [Result] Pichichero M, Papa T, Blatter M, Mitchell D, Kratz R, Sneed J, Bassily E, Casey J, Gilmet G. Immune memory in children previously vaccinated with an experimental quadrivalent meningococcal polysaccharide diphtheria toxoid conjugate vaccine. Pediatr Infect Dis J. 2006 Nov;25(11):995-1000. doi: 10.1097/01.inf.0000243215.46312.4a. PMID 17072120
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 10 march through 13 June 2003 in 8 US clinic sites
Pre-assignment Details: A total of 173 participants that met the inclusion and exclusion criteria were enrolled and vaccinated.
Groups:
- Meningococcal Vaccine-naive: Participants have never received a Meningococcal vaccine in the past.
Period: Overall Study
Arm/Group | Previously Received TetraMenD | Meningococcal Vaccine-naive
Started | 102 | 71
Completed | 100 (Two participants had vaccination errors, they were removed from analysis.) | 61
Not Completed | 2 | 10
Not completed — Lost to Follow-up | 0 | 8
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Vaccination error-wrong dose/expired lot | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Previously Received TetraMenD | Meningococcal Vaccine-naive | Total
Number analyzed (Participants) | 100 | 71 | 171
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 100 | 71 | 171.0
  Between 18 and 65 years | 0 | 0 | 0.0
  >=65 years | 0 | 0 | 0.0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.5 (0.52) | 3.8 (0.87) | 4.2 (0.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 44 | 86.0
  Male | 58 | 27 | 85.0
Region of Enrollment [Number; unit: participants]
  United States | 100 | 71 | 171.0

OUTCOME MEASURES:

1. Other Pre Specified Outcome: Percentage of Participants With at Least a 4-fold Rise in Serum Bactericidal Activity to Each Vaccine Meningococcal Serogroups.
Time Frame: Baseline to Day 8 and Day 28 post-vaccination
Population: Fold rise analysis was assessed in per-protocol population with valid serology data.
Measure: Number; unit: Percentage of participants
Arm/Group | Previously Received TetraMenD | Meningococcal Vaccine-naive
Number analyzed (Participants) | 46 | 35
Percentage of participants
  Meningococcal Serogroup A (Day 8) | 93 | 89
  Meningococcal Serogroup C (Day 8) | 91 | 89
  Meningococcal Serogroup Y (Day 8) | 96 | 74
  Meningococcal Serogroup W-135 (Day 8) | 98 | 100
  Meningococcal Serogroup A (Day 28) | 72 | 85
  Meningococcal Serogroup C (Day 28) | 93 | 54
  Meningococcal Serogroup Y (Day 28) | 78 | 65
  Meningococcal Serogroup W-135 (Day 28) | 93 | 100

2. Other Pre Specified Outcome: Percentage of Participants Reporting Solicited Local and Systemic Reactions Within Days 0 to 7 Post-vaccination.
Time Frame: Day 0 to 7 post-vaccination
Population: Safety analysis was on all enrolled and vaccinated subjects with available reaction data, intent-to-treat population.
Measure: Number; unit: Percentage of participants
Arm/Group | Previously Received TetraMenD | Meningococcal Vaccine-naive
Number analyzed (Participants) | 100 | 69
Percentage of participants
  Any Solicited Local Reaction (Days 0-7) | 46 | 45
  Any Grade 3 Solicited Local Reaction (Days 0-7) | 0 | 0
  Any Redness | 23 | 20
  Grade 3 Redness (>2 inch) | 0 | 0
  Any Swelling | 11 | 15
  Grade 3 Swelling (>2 inch) | 0 | 0
  Any Induration | 14 | 13
  Grade 3 Induration (>2 inch) | 0 | 0
  Any Pain | 34 | 33
  Grade 3 Pain (Disabling, unable to move arm) | 0 | 0
  Any Solicited Systemic Reaction (Days 0-7) | 38 | 42
  Any Grade 3 Solicited Systemic Reaction (Days 0-7) | 3 | 4
  Any Fever | 10 | 3
  Grade 3 Fever (≥ 40.0°C) | 0 | 0
  Any Fussiness | 22 | 30
  Grade 3 Fussiness (Irritability for > 3 hours) | 1 | 1
  Any Drowsiness | 17 | 12
  Grd 3 Drowsiness: not interested in usual activity | 1 | 1
  Any Anorexia | 8 | 13
  Grade 3 Anorexia (Skipped ≥ 3 meals) | 1 | 1
  Any Vomiting | 5 | 0
  Grade 3 Vomiting (≥ 3 episodes) | 2 | 0
  Any Diarrhea | 6 | 9
  Grade 3 Diarrhea (≥ 5 episodes) | 0 | 0

3. Primary Outcome: Geometric Mean Titers (GMT) of Serum Bactericidal Activity for Each Vaccine Serogroups Before and Post-vaccination.
Time Frame: Day 0 and Days 8 and 28 post-vaccination
Population: Geometric mean titers were determined in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Previously Received TetraMenD | Meningococcal Vaccine-naive
Number analyzed (Participants) | 100 | 61
Titers
  Meningococcal Serogroup A (Day 0) | 316.1 [182.6 to 547.2] | 126.5 [67.3 to 237.9]
  Meningococcal Serogroup A (Day 8) | 11411.9 [9196.5 to 14161.1] | 6720.1 [5205.0 to 8676.2]
  Meningococcal Serogroup A (Day 28) | 5620.6 [4321.2 to 7310.8] | 2603.3 [1767.0 to 3835.3]
  Meningococcal Serogroup C (Day 0) | 68.4 [41.2 to 113.6] | 21.2 [11.6 to 38.9]
  Meningococcal Serogroup C (Day 8) | 8700.9 [6185.5 to 12239.1] | 2447.5 [1651.9 to 3626.3]
  Meningococcal Serogroup C (Day 28) | 7261.6 [5213.5 to 10114.4] | 300.4 [128.8 to 700.4]
  Meningococcal Serogroup Y (Day 0) | 411.5 [286.9 to 590.1] | 241.8 [138.3 to 422.9]
  Meningococcal Serogroup Y (Day 8) | 7261.6 [5696.2 to 9257.2] | 3859.7 [2751.1 to 5414.9]
  Meningococcal Serogroup Y (Day 28) | 3798.7 [2735.7 to 5274.8] | 1410.0 [939.9 to 2115.3]
  Meningococcal Serogroup W-135 (Day 0) | 92.5 [57.9 to 147.8] | 17.5 [10.8 to 28.2]
  Meningococcal Serogroup W-135 (Day 8) | 11761.1 [8556.4 to 16166.0] | 5194.8 [3849.3 to 7010.5]
  Meningococcal Serogroup W-135 (Day 28) | 6245.9 [4231.8 to 9218.5] | 2103.3 [1303.7 to 3393.3]

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination to 28 days post-vaccination.
Arm/Group | Previously Received TetraMenD | Meningococcal Vaccine-naive
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/71
Other Adverse Events (participants affected / at risk) | 34/100 | 33/71
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Previously Received TetraMenD (N=100) | Meningococcal Vaccine-naive (N=71)
Injection site erythema (General disorders) | 23 | 20/69
Injection site swelling (General disorders) | 11 | 15/69
Injection site Induration (General disorders) | 14 | 13/69
Injection site pain (General disorders) | 34 | 33/69
Pyrexia (General disorders) | 10 | 3/69
Vomiting NOS (Gastrointestinal disorders) | 5 | 0/69
Somnolence (Nervous system disorders) | 17 | 12/69
Anorexia (Metabolism and nutrition disorders) | 8 | 13/69
Irritability (Psychiatric disorders) | 22 | 30/69
Diarrhoea (Gastrointestinal disorders) | 6 | 9/69
Nasopharyngitis (Infections and infestations) | 3 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.